CLINICAL TRIAL: NCT00108264
Title: Tumor RNA Transfected Dendritic Cell Vaccines
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: CLIN-021-02S
Record Dates: First submitted 2005-04-14; First posted 2005-04-15 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2007-05

CONDITIONS: Prostate Cancer
Keywords: Prostatic Neoplasms; Neoplasm Metastasis; Immunotherapy; Active; Dendritic Cells
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis; Motor Activity

INTERVENTIONS:
Biological: Tumor RNA transfected dendritic cells

SUMMARY:
The purpose of this study is to use dendritic cells transfected with amplified RNA from autologous tumor cells to develop a vaccine strategy for the treatment of prostate cancer in patients with disseminated disease.

DETAILED DESCRIPTION:
The specific aims are: 1) to evaluate, in a phase I clinical trial, the safety of vaccinating patients with dendritic cells transfected with RNA from autologous cancer cells; 2) to analyze the T cell responses induced by the treatment; and 3) to improve the efficacy of the treatment by developing methods to increase the induction of CD4+T cell responses.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histologically confirmed diagnosis of metastatic prostate cancer stages D1 - D3 are eligible for this study.
* They must not have a history of autoimmune disease, serious intercurrent chronic or acute illness, pulmonary disease, active hepatitis, serologic evidence for HIV, or be receiving corticosteroid or immunosuppressive therapy.

Exclusion Criteria:

* Patients will be excluded from the study if they have received chemotherapy or other forms of immunotherapy in the 6 weeks prior to study entry.

Min Age: 10 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Study Completion 2005-09

CONTACTS AND LOCATIONS:
Locations (1):
- Durham VA Medical Center, Durham, North Carolina, United States